CLINICAL TRIAL: NCT01248156
Title: The Maintenance of Human Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 101311; K24HL103800 (NIH)
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intervention: Patients with persistent, long standing persistent and paroxysmal AF, who will receive ablation at sites that potentially maintain human AF.
- Control: Patients with persistent, long standing persistent and paroxysmal AF, who receive conventional ablation as determined by the operator at each site, and based upon Heart Rhythm Society guidelines.

SUMMARY:
Atrial fibrillation (AF) is the most prevalent heart rhythm disorder in the United States, affecting 2.5 million individuals in whom it may cause stroke, palpitations, heart failure, and even death. Unfortunately, therapy for AF is limited. Anti-arrhythmic or rate-controlling drugs are poorly tolerated, with frequent side effects and do not reduce stroke risk. Ablation is an emerging, minimally invasive therapy that has attracted considerable attention because it may eliminate AF. Unfortunately, AF ablation is technically challenging, with a success of only 50-70% (versus >90% for other arrhythmias) and serious risks. A major cause of these limitations is that the mechanisms for human AF are not known and thus ablation cannot be directed to them. As a result, AF ablation is empiric and results in extensive destruction of the atrium.

This project will perform research to better understand AF and determine if abnormal activity in small regions or more widespread regions of the heart cause AF. By performing these studies in patients during clinical procedures, this project may lead to a paradigm shift in the understanding and treatment of AF.

DETAILED DESCRIPTION:
This proposal will test the hypothesis that spatially localized sites maintain ongoing human AF, so that ablation at these drivers may eliminate AF on long-term followup. The investigators will study atrial fibrillation in patients undergoing ablation, to identify regions that may be sustaining AF, then ablate at them.

The study design will be to identify sites that may be maintaining AF, using mapping of AF prior to ablation. Once identified, these sites will be targeted for ablated using traditional methods. This process will be repeated up to six times. The locations of these sites will be recorded, and compared to traditional sites for AF ablation, including the pulmonary veins and left atrial roof. They will also be studied for the presence of complex fractionated electrograms and high dominant frequency.

Patients with persistent, long standing persistent, and paroxysmal AF will be included, and patients will then be followed for 6-12 months.

ELIGIBILITY:
INCLUSION CRITERIA for STUDY SUBJECTS:

* patients undergoing electrophysiology study (EPS) for ablation of (a) paroxysmal AF (non-rheumatic) whose AF episodes self-terminate in < 7 days, or (b) persistent AF (non-rheumatic) whose AF episodes last >or= 7 days but terminate with DC cardioversion or anti-arrhythmic drugs and do not recur within 24 hours.
* AF patients must have failed >or= 1 anti-arrhythmic drug

INCLUSION CRITERIA for ALL SUBJECTS:

* will have a full evaluation focusing on diabetes mellitus, hypertension, coronary disease, left ventricular ejection fraction (LVEF). We will document whether AF relates to times of vagal activity (meals or sleep) or exercise. We will record the use of drugs affecting the renin-aldosterone-angiotensin system (RAAS) and statins, that may protect against atrial fibrosis and AF. We will document serum potassium level, since slight elevations slow CV in vitro. We will record 12-lead ECG and echocardiography for left atrial diameter, and stress test and/or coronary angiography if indicated.
* will have event monitor recordings with daily transmissions for at least one week to document AF burden (study subjects) or exclude AF (control subjects).
* must have with-held amiodarone for > 30 days and other anti-arrhythmic drugs for > 5 half-lives.

EXCLUSION CRITERIA FOR ALL SUBJECTS:

* active coronary ischemia in the past year, since the protocol uses isoproterenol
* rheumatic valve disease, that leads to distinct AF and increases thromboembolic risk
* prior ablation or cardiac surgery, that alters atrial electrophysiology
* LA clot or dense contrast on TEE
* deranged serum electrolytes, and K+ outside 4.0-5.0 mmol/l
* left atrial diameter > 60 mm
* LVEF < 40% or New York Heart Association heart failure > Class II, to exclude distinct, heart-failure related remodeling
* thrombotic disease, venous filters, transient ischemic attack or cerebrovascular accident, to minimize additional risk
* pregnancy, to minimize fluoroscopy. As part of routine clinical care, all female patients of childbearing age receive a ß-HCG pregnancy test. Any who test positive will not be included in the research study
* inability or unwillingness to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be men and women of all races aged above 21 years undergoing clinically indicated ablation of persistent and paroxysmal AF subjects.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
recurrence of atrial fibrillation | 1 year
  recurrence of AF measured using clinical follow-up with implanted devices in all patients who consent

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Narayan, MD, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California San Diego Medical Center, San Diego, California
  - Veterans Affairs San Diego Medical Center, San Diego, California